CLINICAL TRIAL: NCT03721861
Title: Use of Neural Functional Electrical Stimulation for the Recovery of Grasping Movements for Patient With Quadriplegia.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment is finished
Sponsor: Clinique Beau Soleil (Other)
Collaborators: Institut National de la recherche en Informatique et Automatique (Unknown); University Hospital, Montpellier (Other); Mxm-Obelia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2014A0175245
Record Dates: First submitted 2018-10-19; First posted 2018-10-26 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injuries
Keywords: neural stimulation; quadriplegia; grasping
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intra-operative neural cuff stimulation — A feasibility study consists of placing 2 electrodes around the radial or medial nerves intraoperatively. The movements caused by the electrical stimulation of these nerves are observed.

SUMMARY:
Functional electrical stimulation (FES) has been used for decades in rehabilitation centers. Having demonstrated efficacy for prevention of muscle atrophy following spinal cord injury (SCI), FES can also be considered for functional restoration of hand movements in the patients with complete tetraplegia belonging to group 0 or 1 of the classification of Giens. However, the majority of the systems using the FES directly stimulates the muscles (surface electrodes, intramuscular or epimysial), which increases the number of components and requires more electrical energy for the muscle activation. Nerve stimulation would activate more muscles through a reduced number of electrodes, limiting the number of internal components, reduces the risk of spreading infections and require less electrical energy for its operation.

ELIGIBILITY:
Inclusion Criteria:

1. Neurological level ≥ C7
2. 18 years old min and max 65 years old,
3. Complete traumatic injury: defined by A or B score on the AIS scale.
4. patient belonging to group 0 or 1 of the Giens classification.
5. neurological stability (no change in muscle testing)> 6 months,
6. post-injury duration> 6 months
7. Patients undergoing surgery to restore elbow extension.
8. threshold of stimulation and diffusion of the studied muscles below 50 mA of intensity for a pulse width of 300 μs and a frequency of 25 Hz.
9. positive electrical mapping of muscles with a minimum score of 4 MRC for at least one of the extensors (triceps, ECRL, ECRB, EDC, EPL) and / or flexor (FPL, FDS, FDP).

Exclusion Criteria:

* 1. strong spasticity and contractures in flexion or extension of the upper limbs.

  2. Unstable epilepsy. 3. Unstable cardiovascular pathology (coronary heart disease, major hypertension, heart failure etc.).

  4. wearing a pacemaker. 5. Dermatological problems contraindicate the application of surface electrodes.

  6. body weight> 100kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-09 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Selectivity of stimulation | a week
  Electrical stimulation of the median or radial nerve via multipolar "cuff" electrodes induces electromyographic signals on a number of muscles.
  If at least 92% of cases, it is possible to selectively stimulate 4 muscle groups (the elbow extensor: triceps, the extensors of the fingers and carp: ECRL, ECRB, EDP, EPL, the flexor of the thumb: FPL and flexors of 4 fingers (II to V): FDS and FDP) to restore 4 functions (elbow, wrist and finger extensions; the 4 fingers and the thumb flexions).
  An activation of a muscle group is considered selective if both the selectivity index is ≥ 0.7 and the recruitment is ≥20%. Finally, there will be success the selective activation induces the right movements (extension of the elbow, extension of the wrist and fingers, flexion of the 4 fingers and flexion of the thumb). There will be failure otherwise.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Beau Soleil, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tigra W, Dali M, William L, Fattal C, Gelis A, Divoux JL, Coulet B, Teissier J, Guiraud D, Azevedo Coste C. Selective neural electrical stimulation restores hand and forearm movements in individuals with complete tetraplegia. J Neuroeng Rehabil. 2020 May 19;17(1):66. doi: 10.1186/s12984-020-00676-4. PMID 32429963